CLINICAL TRIAL: NCT07069595
Title: PREDICT-RD: Postoperative Molecular Residual Disease by ctDNA Surveillance in TNBC With Residual Disease
Brief Title: PREDICT-RD: ctDNA Surveillance in TNBC With Residual Disease
Acronym: PREDICT-RD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: AstraZeneca (Industry); Translational Breast Cancer Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2215
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Residual Disease; Triple Negative Breast Cancer (TNBC); Stage II/III
Keywords: circulating tumor DNA (ctDNA); surveillance; Dato-DXd
MeSH Terms: conditions — Breast Neoplasms; Neoplasm, Residual; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Patients with higher residual cancer burden (Experimental): Participants with stage II/III triple negative breast cancer (TNBC) and residual disease post-neoadjuvant therapy, particularly patients with higher residual cancer burden (RCB II/III), remain at high risk for developing recurrence.
  Interventions: Drug: Datopotamab deruxtecan; Diagnostic Test: Circulating tumor DNA (ctDNA) testing

INTERVENTIONS:
Drug: Datopotamab deruxtecan — Dato-DXd is administered adjuvantly at 6 mg/kg IV for eight cycles.
  Other Names: Dato-DXd
Diagnostic Test: Circulating tumor DNA (ctDNA) testing — Circulating tumor DNA (ctDNA) testing is a type of biopsy that analyzes fragments of DNA shed by cancer cells into the bloodstream. These fragments, known as ctDNA, can provide valuable information about the genetic makeup of a tumor without needing a traditional tissue biopsy.

SUMMARY:
This is a Phase II, interventional, prospective, single-arm, multi-center study that will enroll patients with stage II/III triple negative breast cancer (TNBC) who have residual cancer burden (RCB) II/III after conventional neoadjuvant chemo-immunotherapy followed by surgery. Technological advances in ctDNA assays have improved both the sensitivity and reliability of molecular residual disease (MRD) detection to enable real-time measurement with clinical-grade assays.

The primary objective of this study will be to evaluate ctDNA-based MRD status in high-risk, early-stage TNBC patients by defining the proportion of TNBC patients with MRD-only recurrence (ctDNA positive without radiographically measurable recurrence) during post-surgery surveillance. The secondary objectives will evaluate the safety, preliminary efficacy, and survival outcomes of using Dato-DXd in participants with MRD-only TNBC.

Dato-DXd is an investigational antibody-drug conjugate (monoclonal antibody specific for TROP2 and a topoisomerase I (Topo-1) inhibitor) that has demonstrated promising efficacy in TNBC patients with a manageable safety profile.

DETAILED DESCRIPTION:
Despite treatment advances, patients with II/III triple negative breast cancer (TNBC) residual disease post-neoadjuvant therapy, particularly patients with higher residual cancer burden (RCB II/III), remain at high risk for developing recurrence. Furthermore, early detection of relapse risk, when the residual disease burden is micrometastatic (defined here as undetectable by standard cross-sectional imaging), provides a chance for disease eradication whereas macrometastatic disease (i.e., detectable on standard cross-sectional imaging) is generally considered to be non-curable.

There are no standard of care (SOC) surveillance strategies for early detection of micrometastatic disease in high-risk TNBC beyond clinical monitoring. Detecting molecular residual disease (MRD) is a promising approach to identifying patients at increased risk of recurrence after definitive therapy, who may benefit from the escalation of their treatment and remain potentially curable with effective systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent was obtained to participate in the study, and HIPAA authorization for the release of personal health information.

* Participant is willing and able to comply with study procedures based on the judgment of the investigator.
* Age ≥ 18 years at the time of consent.
* Histological confirmation of TNBC defined by ER/PR <10%, HER2 0-1+ by IHC or 2+ by IHC and fluorescence in situ hybridization (FISH) negative.
* Stage II/III TNBC treated with neoadjuvant systemic therapy AND have residual disease defined as RCB II/III at time of surgery.
* Baseline staging scans at the discretion of the treating physician and demonstrate no evidence of metastatic disease.
* The participant must have archival diagnostic tissue and/or surgical resection tissue Available.
* Participants are willing and able to comply with study procedures based on the judgment of the investigator.

Exclusion Criteria:

• Participants are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
The proportion of triple negative breast cancer (TNBC) with molecular residual disease (MRD) | Up to 3 years after registration
  The number of participants with triple negative breast cancer (TNBC) with molecular residual disease (MRD) only recurrence, which is defined as ctDNA positivity without radiographically measurable recurrence, during post-surgery surveillance.

SECONDARY OUTCOMES:
The time between Circulating tumor DNA (ctDNA) positivity and clinically proven relapse | Up to 3 years after registration
  ctDNA levels will be measured every 6 weeks during adjuvant and/or Dato-DXd therapy and every 12 weeks thereafter.
Duration of Circulating tumor DNA (ctDNA) clearance | Up to 3 years after registration
  Duration of ctDNA clearance will be defined as the time from the first confirmed clearance (for negative test after positive results) to the date of confirmed positivity.
Circulating tumor DNA (ctDNA) clearance with Dato-DXd | Up to 3 years after registration
  ctDNA clearance in participants who receive Dato-DXd will be defined as the proportion of participants who convert from ctDNA positive to negative after initiation of Dato-DXd.
Toxicity of Dato-DXd | Up to 3 years after registration
  Toxicity of Dato-DXd treatment will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. NCI-CTCAE is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Recurrence Free Survival (RFS) for ctDNA-positive and ctDNA-negative disease. | Up to 3 years after registration
  RFS will be measured from the day of the first circulating tumor DNA (ctDNA) measurement to documented recurrence of disease in participants with ctDNA-positive and ctDNA-negative disease.
Recurrence Free Survival (RFS) - Dato-DXd | Up to 3 years after registration
  RFS will be measured from the day of the first circulating tumor DNA (ctDNA) measurement to documented recurrence of disease in participants who receive Dato-DXd.
Overall Survival (OS) - ctDNA-positive and ctDNA and negative disease. | Up to 3 years after registration
  OS will be measured from the day of the first ctDNA measurement to death from any cause in participants with ctDNA-positive and ctDNA-negative disease.
Overall Survival (OS) - for ctDNA-positive and ctDNA-negative disease. | Up to 3 years after registration
  OS will be measured from the day of the first ctDNA measurement to death from any cause in participants who receive Dato-DXd.

CONTACTS AND LOCATIONS:
Overall Officials: Yara Abdou, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials